CLINICAL TRIAL: NCT02208908
Title: Oral Care and Cancer: Assessing the Contribution of Training Healthcare Teams to Support the Oral Status of Patients Hospitalized in Palliative Situation
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: BBC3
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Management of Oral Care and Cancer in Palliative Situation
Keywords: Oral care; cancer; palliative; training
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patient with cancer hospitalize inpalliative situation: An accurate assessment of the oral condition and proper care will be carried out on day 2 (J2) of hospitalization and repeated on the day of hospital discharge by the nurse detached service, regardless of caregivers.
  An assessment of the traceability of clinical assessment and appropriate treatment prescribed or will be conducted on day 3 and repeated the day of the release of hospitalization (or day 15) from information recorded in the patient record
  Interventions: Other: Evaluation of the oral conditionand proper care

INTERVENTIONS:
Other: Evaluation of the oral conditionand proper care — An accurate assessment of the oral condition and proper care will be carried out on day 2 (J2) of hospitalization and repeated on the day of hospital discharge by the nurse detached service, regardless of caregivers.

SUMMARY:
The purpose of this study is to measure the impact of training on the practical assessment and management of the oral status of patients hospitalized in palliative situation.

DETAILED DESCRIPTION:
According to the French support and palliative care (RFS) Company, palliative care are active in a holistic approach to the person with a serious illness, progressive or terminal. Their goal is to relieve physical symptoms and other pain and take into account the psychological, social and spiritual suffering.

He consensus among caregivers to recognize the importance and maintaining good oral hygiene for patients treated for cancer at all ages of life, home and in hospital, and consider that the oral hygiene is an integral part of nursing, toilet and contributes to the health of patients. This is primarily a comfort for the person to have a healthy mouth, healthy with a clean mouth, but also a tool that meets all its features.

The feeding, respiration and communication are three closely related to the proper functioning of the oral cavity needs. Furthermore, cancer, various treatments, age are possible disturbances oral integrity. The nurse helped the caregiver has upstream of care, the role of counseling and prevention. However, a review of the oral and / or the establishment of procedures support oral hygiene status are largely neglected despite the existence of published recommendations. This is particularly related to lack of information provided and continuing education offered to carers and the lack of written procedures. Moreover, the limited literature on the subject limit the possibility of initiatives, the establishment of a procedure before relying on evidence-based practice. Measure 43 Cancer Plan I and the establishment of mobile units or palliative care teams and management of pain in Residential Care (especially CHU and Centres for the Fight Against Cancer [PBC] ) is an opportunity to implement an audit action.

This project is part of a research program in several steps. From November 2010 to August 2011, 260 patients (107 hommes/153 women), median age 64 years (19-88 years) were included. J2, a healthy mouth, moderately (dry mouth and / or dirty) or severely (fungal mouth and / or painful ulcerated and / or hemorrhagic) was altered respectively observed for 61 (23.5%), 139 (53.5%) and 60 (23.0%) patients. Traceability of this oral assessment is found in 10% of cases. The exit assessment was performed in 184 patients (46 deaths, 30 non-assessed), including 129 with a delay ≥ 5 days between J2 and output. The mouth on the output shows a healthy mouth, moderately and severely impaired in 33 (26%), 70 (54%) and 26 (20%) of these 129 patients, respectively. Thus, 27 (21%) patients showed deterioration in their oral condition during hospitalization: 13/31 (42%) for patients with a healthy mouth to J2 and 14/72 (19%) for those with a mouth moderately altered to J2. In contrast, 28/129 (22%) patients, including 13/72 (18%) and 15/26 (58%) respectively had a mouth moderately and severely impaired the initial assessment have improved access to oral output state .

Following this audit action, a tool Medical Assessment mouth has been prepared in collaboration with health care teams participating as well as recommendations for management of each type of mouth (concerning both hygiene as drug and non-drug measures), in agreement with those of learned societies, a plan of care by type of mouth care.

An inter centers presenting the results of the first stage (inventory) and definition of the training plan was held in March 2013 in the presence, for each center, doctor, and nurse care manager and / or scope of health involved in palliative care and research program. The purpose of this meeting was to present the evaluation grid of mouth and recommendations developed state care and the plan and tools for training healthcare teams on site.

From May to September 2013, personnel, formed during this meeting, provide training for paramedical and medical teams of their establishment.

The purpose of this study is to measure the impact of training on the practical assessment and management of the oral status of patients hospitalized in palliative situation.

Expected results We hope that the appropriate training of health care teams allow all patients during their hospitalization benefit systematically evaluate the oral condition, the implementation of actions consistent with the recommendations and thus an improvement the care of their oral condition.

Ultimately, it is hoped that the management of the oral condition falls within the overall care of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years with cancer and palliative hospital situation
* Patient able to communicate with the nursing staff;
* Patient able to understand the meaning of the questions;
* Patients whose length of stay is at least 5 days
* Patients whose life expectancy is greater than or equal to three weeks;
* Patients who have given their written consent to the study participation.

Exclusion Criteria:

* Patient refusing to make the clinical assessment;
* Patient not giving their consent for participation;
* Patient unable to communicate with the nursing staff;
* Patient not proficient in the French language;
* Patient suffering from cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cancer hospitalize inpalliative situation
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an improvement of 10% of the buccal state | up to day 15

SECONDARY OUTCOMES:
The quality and adequacy of the prescription (non-drug and / or drug attitudes) to record oral | Day 2 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine GRACH, MD, Principal Investigator — Centre François Baclesse
Locations (5):
- France (5):
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre François Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Henri Becquerel, Rouen